CLINICAL TRIAL: NCT02649634
Title: Adding Motivational Interviewing to a Behavioral Weight Loss Treatment for Obesity: A Randomized Controlled Trial
Brief Title: Does Motivational Interviewing Improve Behavioral Weight Loss Outcomes for Obesity?
Acronym: BWLP+MI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Kristin von Ranson, Associate Professor, Psychology, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CFREB#5297
Record Dates: First submitted 2016-01-05; First posted 2016-01-07 (Estimated); Results first posted 2017-03-20 (Actual); Last update posted 2017-03-20 (Actual); Status verified 2017-01

CONDITIONS: Obesity; Overweight
Keywords: Motivational Interviewing; Obesity; Weight Loss; Behavioral Medicine
MeSH Terms: conditions — Obesity; Overweight; Weight Loss | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motivational Interviewing (Experimental): Two 45-60 minute motivational interviewing sessions focusing on exploring and resolving ambivalence towards change.
  Interventions: Behavioral: Motivational Interviewing
- Attention Control (Active Comparator): Two 45-60 minute semi-structured interviews, acting as a pseudo-intervention, ascertaining information relevant to health history, weight history, diet history, as well as dietary and physical activity habits.
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: Motivational Interviewing — The semi-structured MI protocol was a 45-60 minute intervention based on general MI principles and guidelines, MI strategies specific to health care practice, and MI principles for obesity treatment. The MI protocol included the following components: (1) eliciting concerns about weight; (2) exploring ambivalence; (3) assessing importance and confidence for change; (4) writing a decisional balance; (5) bolstering self-efficacy; (6) looking towards the future; and (8) eliciting ideas for possible changes participant could make to work towards weight loss. Although there was slight variation, the protocol for both MI sessions consisted of similar components.
  Arms: Motivational Interviewing
Behavioral: Attention Control — The attention control interview was a semi-structured interview ascertaining information relevant to health history, weight history, diet history, dietary and physical activity habits. The majority of questions for the control interviews were drawn from the Behavioural Weight Loss Program intake application. It was designed to be structurally equivalent to the MI session in terms of length of session, timing of sessions, and treatment modality. The goal of the attention-control interview was to provide a pseudo-intervention that controlled for factors common to attending treatment (e.g., attending treatment sessions, having personal contact with a therapist, discussing weight-related issues).
  Arms: Attention Control

SUMMARY:
The purpose of this study is to determine whether adding motivational interviewing (MI) to a behavioural weight loss program (BWLP) results in improved weight loss for adults who are overweight or obese.

DETAILED DESCRIPTION:
Although behavioural weight loss programs (BWLP) are typically the first line of treatment for obesity, they are often plagued by high attrition rates and poor adherence. Studies evaluating the benefit of adding motivational interviewing (MI) to BWLPs have yielded mixed findings. The main purpose of this randomized controlled trial was to assess the efficacy of adding MI to a BWLP on weight loss and adherence outcomes among 135 overweight and obese individuals enrolled in a 12-week (24 session) BWLP.

This study used a randomized, controlled, longitudinal, between-subjects design to investigate the effects of a two-session MI intervention on weight loss in participants enrolled in a BWLP. Patients received either two 45-60 minute MI interventions or two 45-60 minute attention control interviews. The control group interview consisted of questions ascertaining weight history, diet history, dietary awareness and physical activity. Questions for the control group focused primarily on assessment of past behaviour whereas questions for the MI group focused on enhancing motivation by exploring and resolving ambivalence. Weight was measured at baseline, end of the BWLP, and 6 months following BWLP completion. Program adherence (measured as number of BWLP sessions attended out of 24) was assessed as a secondary dependent measure. Importance, readiness, and confidence for weight change were assessed at baseline and then immediately following each interview (either MI or control). In addition, several other secondary outcome measures were assessed at baseline, end of the BWLP, 1 month follow-up, and 6 month follow-up.

Research personnel informed all BWLP participants about the study at the initial BWLP group intake assessments, which occurred just prior to the commencement of the formal BWLP. Individuals who expressed interest in participating were contacted by phone by a research assistant and screened for eligibility. If eligible, an appointment was made for the first MI/control session which was scheduled within the first two weeks of the BWLP. Randomization occurred immediately prior to this interview. Participants were then contacted during the 10th week of the BWLP to schedule a second MI/control session, which occurred approximately during the 12th week of the program. Participants were all contacted several weeks following program completion to schedule the one-month follow-up assessment. Finally, all participants were contacted approximately five months following program completion in order to schedule the six-month follow-up assessment.

Sessions were tape recorded for all participants for quality assurance purposes. A subset of tapes were used to assess for treatment integrity.

ELIGIBILITY:
Inclusion Criteria:

* Overweight to obese (BMI greater than or equal to 25 kilograms per meter squared).

Exclusion Criteria:

* Pregnancy (or intention of becoming pregnant within 9 months)
* Health issues that would preclude participation in physical activity
* Concurrent involvement in another weight loss program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2007-09; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin M von Ranson, PhD, Principal Investigator — University of Calgary

IPD SHARING:
Plan to Share IPD: Yes
Data uploaded to Zenodo.org

REFERENCES:
- [Background] Armstrong MJ, Mottershead TA, Ronksley PE, Sigal RJ, Campbell TS, Hemmelgarn BR. Motivational interviewing to improve weight loss in overweight and/or obese patients: a systematic review and meta-analysis of randomized controlled trials. Obes Rev. 2011 Sep;12(9):709-23. doi: 10.1111/j.1467-789X.2011.00892.x. Epub 2011 Jun 21. PMID 21692966
- [Background] West DS, DiLillo V, Bursac Z, Gore SA, Greene PG. Motivational interviewing improves weight loss in women with type 2 diabetes. Diabetes Care. 2007 May;30(5):1081-7. doi: 10.2337/dc06-1966. Epub 2007 Mar 2. PMID 17337504
- [Background] DiMarco ID, Klein DA, Clark VL, Wilson GT. The use of motivational interviewing techniques to enhance the efficacy of guided self-help behavioral weight loss treatment. Eat Behav. 2009 Apr;10(2):134-6. doi: 10.1016/j.eatbeh.2009.02.001. Epub 2009 Feb 15. PMID 19447358
- [Background] Webber KH, Gabriele JM, Tate DF, Dignan MB. The effect of a motivational intervention on weight loss is moderated by level of baseline controlled motivation. Int J Behav Nutr Phys Act. 2010 Jan 22;7:4. doi: 10.1186/1479-5868-7-4. PMID 20157441
- [Background] DiLillo V, Siegfried NJ, West DS. Incorporating motivational interviewing into behavioral obesity treatment. Cognitive and Behavioral Practice 10(2): 120-130, 2003.
- [Background] Hemmelgarn BR, McAlister FA, Grover S, Myers MG, McKay DW, Bolli P, Abbott C, Schiffrin EL, Honos G, Burgess E, Mann K, Wilson T, Penner B, Tremblay G, Milot A, Chockalingam A, Touyz RM, Tobe SW; Canadian Hypertension Education Program. The 2006 Canadian Hypertension Education Program recommendations for the management of hypertension: Part I--Blood pressure measurement, diagnosis and assessment of risk. Can J Cardiol. 2006 May 15;22(7):573-81. doi: 10.1016/s0828-282x(06)70279-3. PMID 16755312
- [Background] Fairburn CG, Beglin SJ. Assessment of eating disorders: interview or self-report questionnaire? Int J Eat Disord. 1994 Dec;16(4):363-70. PMID 7866415
- [Background] Paffenbarger RS Jr, Wing AL, Hyde RT. Physical activity as an index of heart attack risk in college alumni. Am J Epidemiol. 1978 Sep;108(3):161-75. doi: 10.1093/oxfordjournals.aje.a112608. PMID 707484
- [Background] Kristal AR, Shattuck AL, Henry HJ. Patterns of dietary behavior associated with selecting diets low in fat: reliability and validity of a behavioral approach to dietary assessment. J Am Diet Assoc. 1990 Feb;90(2):214-20. PMID 2303658
- [Background] Clark MM, Abrams DB, Niaura RS, Eaton CA, Rossi JS. Self-efficacy in weight management. J Consult Clin Psychol. 1991 Oct;59(5):739-44. doi: 10.1037//0022-006x.59.5.739. PMID 1955608
- [Derived] Moss EL, Tobin LN, Campbell TS, von Ranson KM. Behavioral weight-loss treatment plus motivational interviewing versus attention control: lessons learned from a randomized controlled trial. Trials. 2017 Jul 25;18(1):351. doi: 10.1186/s13063-017-2094-1. PMID 28743313

RESULTS

PARTICIPANT FLOW:
Groups:
- Motivational Interviewing: Two 45-60 minute motivational interviewing sessions focusing on ambivalence towards change.
  Motivational Interviewing: The semi-structured MI protocol was a 45-minute intervention based on general MI principles and guidelines, MI strategies specific to health care practice, and MI principles for obesity treatment. The MI protocol included the following components: (1) eliciting concerns about weight; (2) exploring ambivalence; (3) assessing importance and confidence for change; (4) writing a decisional balance; (5) bolstering self-efficacy; (6) looking towards the future; and (8) eliciting ideas for possible changes participant could make to work towards weight loss. Although there was slight variation, the protocol for both MI sessions consisted of similar components.
- Attention Control: Two 45-60 minute semi-structured interviews ascertaining information relevant to health history, weight history, diet history, dietary and physical activity habits, acting as a pseudo-intervention.
  Attention Control: The attention control interview was a semi-structured interview ascertaining information relevant to health history, weight history, diet history, dietary and physical activity habits. The majority of questions for the control interviews were drawn from the Behavioural Weight Loss Program intake application. It was designed to be structurally equivalent to the MI session in terms of length of session, timing of sessions, and treatment modality. The goal of the attention-control interview was to provide a pseudo-intervention that controlled for factors common to attending treatment (e.g., attending treatment sessions, having personal contact with a therapist, discussing weight-related issues).
Period: Overall Study
Arm/Group | Motivational Interviewing | Attention Control
Started | 69 | 66
Completed | 66 | 60
Not Completed | 3 | 6
Not completed — Withdrawal by Subject | 3 | 5
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Motivational Interviewing | Attention Control | Total
Number analyzed (Participants) | 69 | 66 | 135
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.56 (9.78) | 44.67 (12.91) | 45.16 (11.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 53 | 105
  Male | 17 | 13 | 30
Region of Enrollment [Number; unit: participants]
  Canada | 69 | 66 | 135
Weight [Mean (Standard Deviation); unit: kilograms] | 95.11 (21.45) | 90.34 (19.46) | 92.78 (20.57)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 33.78 (5.98) | 33.37 (6.58) | 33.58 (6.26)
Physical Activity (PPAQ) [Mean (Standard Deviation); unit: kilocalories per week] — The Paffenbarger questionnaire (PPAQ) assesses amount of planned and lifestyle associated physical activity performed during a typical week. The PPAQ consists of three components: (1) stair climbing, (2) walking, and (3) sports and recreation. Participants report the frequency and duration of physical activity in the past week. Scoring yields energy expenditure from physical activity per week (kcal/kg/week). Higher scores translate into greater energy expenditure per week (i.e.,better outcome). Range is 0 - no theoretical maximum. Highest observed score in our study was 10902 kcal/kg/week.
  kilocalories per week | 1574.46 (1284.43) | 1183.37 (1106.95) | 1384.93 (1213.04)
Dietary Behaviour (DHQ) - overall score [Mean (Standard Deviation); unit: units on a scale] — The Fat-related Dietary Habits Questionnaire (DHQ) is a 22-item questionnaire that was used to collect information on dietary behaviours and high-fat eating patterns. The DHQ consists of an overall summary score and five subscale scores assessing different dimensions of fat-related dietary habits. The overall summary score is the mean of all non-missing subscales scores. Responses are scored on a 4-point scale (usually, often, sometimes, rarely/never). Range of overall summary score is 1 - 4. Higher scores correspond to higher fat intakes (i.e., higher scores = worse outcome).
  units on a scale | 2.90 (0.47) | 2.78 (0.44) | 2.84 (0.46)
Blood Pressure [Mean (Standard Deviation); unit: mmHg]
  Systolic | 129 (13.52) | 129 (13.46) | 129 (13.44)
  Diastolic | 78 (9.77) | 78 (10.66) | 78 (10.18)
Eating Disorder Symptomology (EDEQ) - global score [Mean (Standard Deviation); unit: units on a scale] — Measured by the Eating Disorder Examination Questionnaire (EDEQ). The EDEQ is a 36-item self-report rating scale, which assesses the presence and degree of specific psychopathology associated with eating disorders over the previous 28 days. Consists of a global score as well as four subscales: Eating Concern, Restraint, Shape Concern, and Weight Concern. The global score is obtained by summing the subscale scores and then dividing this sum by the number of subscales (i.e. four). Range is 0 - 6. Higher scores are indicative of greater eating disorder symptomatology (i.e., worse outcome).
  units on a scale | 2.27 (1.08) | 2.34 (0.90) | 2.30 (0.99)
Self-efficacy for Engaging in Physical Activity (ESE) [Mean (Standard Deviation); unit: units on a scale] — The Exercise Self-Efficacy Scale (ESE), is a six-item measure that assessed self-efficacy for engaging in physical activity. Participants rated their confidence that they could exercise on a 5-point Likert scale for six barriers to exercise (e.g., bad weather, stress, availability of equipment). Scores range from 1 - 5. Higher scores are indicative of greater self-efficacy (i.e., higher scores = better outcome).
  units on a scale | 2.84 (0.81) | 2.83 (0.88) | 2.84 (0.84)
Self-efficacy Related to Eating Patterns (WEL) - global score [Mean (Standard Deviation); unit: units on a scale] — The Weight Efficacy Lifestyle Questionnaire (WEL) is a 20-item measure that yields 5 subscale scores which rate self-efficacy for controlling eating in different dimensions: negative emotions, availability, social pressure, physical discomfort, and positive activities. A global/total score (which ranges from 0 - 180) is obtained by summing the scores of each of the five subscales. Higher scores are indicative of greater self-efficacy (i.e., higher scores = better outcome).
  units on a scale | 121.68 (31.63) | 117.87 (33.79) | 119.82 (32.63)

OUTCOME MEASURES:

1. Primary Outcome: Weight at End of Behavioural Weight Loss Program, 12 Weeks
Description: Weight was measured to the nearest 0.1 kg using a balance beam scale
Time Frame: Mean weight recorded at the end of the behavioural weight loss program (week 12)
Population: The participant numbers above represent the number of people that were analyzed on this specific outcome measure, which varies outcome to outcome, and does not necessarily match the number of participants that completed interviews at various stages as listed in the Participant Flow Module.
Measure: Mean (Standard Error); unit: kilograms
Arm/Group | Motivational Interviewing | Attention Control
Number analyzed (Participants) | 64 | 65
kilograms | 89.02 (.43) | 90.09 (.45)
Statistical Analysis 1: Comparison: Motivational Interviewing vs Attention Control; Linear mixed modelling (LMM) was used; Test type: Non-Inferiority or Equivalence — Estimated sample size needed was 90 (45/group). This was based on a sample size calculation for 2 groups with 0.05 alpha, 0.80 power, anticipating a medium effect size (most recent meta-analysis on efficacy of MI on dietary behaviours yielded a medium effect size of .53; Burke et al., 2003). Additionally, for MLM, estimates involving the Level 2 variable (i.e., participants) require samples larger than 50 (Maas & Hox, 2005). Others have suggested 30-50 participants (Scherbaum & Ferreter, 2009); p > .05, Mixed Models Analysis — Significance threshold is p=.05

2. Secondary Outcome: Weight at 6 Month Follow up
Description: a digital scale (Tanita BWB-800S), which assessed weight to the nearest 0.1 kg, was used for the 6 month follow-up assessment
Time Frame: Mean weight 6 months after the end of the behavioural weight loss program
Population: as for outcome 1
Measure: Mean (Standard Error); unit: kilograms
Arm/Group | Motivational Interviewing | Attention Control
Number analyzed (Participants) | 65 | 59
kilograms | 91.26 (.42) | 91.59 (.45)
Statistical Analysis 1: Comparison: Motivational Interviewing vs Attention Control; Linear Mixed Modelling (LMM) was used; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p > .05, Mixed Models Analysis — Significance threshold is p=.05

3. Secondary Outcome: Adherence
Description: The mean number of missed behavioural weight loss sessions (out of 24 sessions)
Time Frame: Assessed once at the end of the behavioural weight loss program (week 12)
Measure: Mean (Standard Deviation); unit: number of group sessions
Arm/Group | Motivational Interviewing | Attention Control
Number analyzed (Participants) | 69 | 66
number of group sessions | 3.71 (4.12) | 4.07 (3.60)
Statistical Analysis 1: Comparison: Motivational Interviewing vs Attention Control; Treatment adherence was analyzed via an independent sample t-test comparing the groups on mean number of TrymGym sessions missed; Test type: Non-Inferiority or Equivalence — Estimated sample size needed was 90 (45/group). This was based on a sample size calculation for 2 groups with 0.05 alpha, 0.80 power, anticipating a medium effect size; p = .65, t-test, 2 sided

4. Secondary Outcome: BMI at End of Behavioural Weight Loss Program, Week 12
Description: Weight was measured to the nearest 0.1 kg using a balance beam scale, height was measured to the nearest 0.1 cm using a stadiometer at the beginning of the behavioural weight loss program. BMI was calculated as weight in Kilograms divided by height in meters squared.
Time Frame: Mean BMI at the end of the behavioural weight loss program (week 12)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: kg/m2
Arm/Group | Motivational Interviewing | Attention Control
Number analyzed (Participants) | 64 | 65
kg/m2 | 32.27 (.16) | 32.64 (.16)
Statistical Analysis 1: Comparison: Motivational Interviewing vs Attention Control; Linear Mixed Modelling (LMM) was used; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p > .05, Mixed Models Analysis — Significance threshold is p=.05

5. Secondary Outcome: BMI at 6 Month Follow up
Description: A digital scale (Tanita BWB-800S), which assessed weight to the nearest 0.1 kg, was used to assess weight for the 6 month follow up assessment, and the height measured at the beginning of the behavioural weight loss program was used to calculate BMI. BMI was calculated as weight in Kilograms divided by height in meter squared.
Time Frame: Mean BMI 6 months after the end of the behavioural weight loss program
Population: as for outcome 1
Measure: Mean (Standard Error); unit: kg/m2
Arm/Group | Motivational Interviewing | Attention Control
Number analyzed (Participants) | 65 | 59
kg/m2 | 32.96 (.16) | 33.11 (.16)
Statistical Analysis 1: Comparison: Motivational Interviewing vs Attention Control; Linear Mixed Modelling (LMM) was used; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p > .05, Mixed Models Analysis — Significance threshold is p=.05

6. Secondary Outcome: Physical Activity at End of the Behavioural Weight Loss Program, Week 12
Description: Physical activity was measured by the Paffenbarger questionnaire (PPAQ; Paffenbarger, Wing, & Hyde, 1978). This self-report questionnaire assesses amount of activity performed during a typical week, and consists of three components: (1) stair climbing, (2) walking, and (3) sports and recreation. Participants were asked to report the frequency and duration of physical activity in the past week. Participants report the frequency and duration of physical activity in the past week. Scoring yields energy expenditure from physical activity per week (kcal/kg/week). Higher scores translate into greater energy expenditure per week (i.e.,better outcome). Range is 0 - no theoretical maximum. Highest observed score in our study was 10902 kcal/kg/week.
Time Frame: Mean physical activity as measured by the PPAQ, at the end of the behavioural weight loss program (week 12)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: kilocalories per week
Arm/Group | Motivational Interviewing | Attention Control
Number analyzed (Participants) | 59 | 59
kilocalories per week | 2161.80 (179.58) | 2211.87 (186.56)
Statistical Analysis 1: Comparison: Motivational Interviewing vs Attention Control; Linear Mixed Modelling (LMM) was used; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p > .05, Mixed Models Analysis — Significance threshold is p=.05

7. Secondary Outcome: Physical Activity at 1 Month Follow up
Description: as for outcome 6
Time Frame: Mean physical activity as measured by the PPAQ, 1 month after the end of the behavioural weight loss program
Population: as for outcome 1
Measure: Mean (Standard Error); unit: kilocalories per week
Arm/Group | Motivational Interviewing | Attention Control
Number analyzed (Participants) | 59 | 52
kilocalories per week | 2196.78 (184.44) | 2299.22 (191.69)
Statistical Analysis 1: Comparison: Motivational Interviewing vs Attention Control; Linear Mixed Modelling (LMM) was used; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p > .05, Mixed Models Analysis — Significance threshold is p=.05

8. Secondary Outcome: Physical Activity at 6 Month Follow up
Description: as for outcome 6
Time Frame: Mean physical activity as measured by the PPAQ, 6 months after the end of the behavioural weight loss program
Population: as for outcome 1
Measure: Mean (Standard Error); unit: kilocalories per week
Arm/Group | Motivational Interviewing | Attention Control
Number analyzed (Participants) | 60 | 55
kilocalories per week | 2060.09 (178.15) | 1789.34 (187.92)
Statistical Analysis 1: Comparison: Motivational Interviewing vs Attention Control; Linear Mixed Modelling (LMM) was used; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p > .05, Mixed Models Analysis — Significance threshold is p=.05

9. Secondary Outcome: Dietary Behaviour at End of the Behavioural Weight Loss Program, Week 12
Description: Dietary behaviour was measured by the Fat-related Dietary Habits Questionnaire (DHQ; Kristal, Shattuck, & Henry, 1990). This self-report questionnaire assesses dietary behaviours and high-fat eating patterns and consists of an overall summary score and five subscale scores assessing different dimensions of fat-related dietary habits. The DHQ consists of an overall summary score and five subscale scores assessing different dimensions of fat-related dietary habits. The overall summary score is the mean of all non-missing subscales scores. Responses are scored on a 4-point scale (usually, often, sometimes, rarely/never). Range of overall summary score is 1 - 4. Higher scores correspond to higher fat intakes (i.e., higher scores = worse outcome).
Time Frame: Mean dietary behaviour score as measured by the overall DHQ score, at the end of the behavioural weight loss program (week 12)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: overall score on DHQ
Arm/Group | Motivational Interviewing | Attention Control
Number analyzed (Participants) | 60 | 60
overall score on DHQ | 2.64 (.04) | 2.62 (.04)
Statistical Analysis 1: Comparison: Motivational Interviewing vs Attention Control; Linear Mixed Modelling (LMM) was used; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p > .05, Mixed Models Analysis — Significance threshold is p=.05

10. Secondary Outcome: Dietary Behaviour at 1 Month Follow up
Description: as for outcome 9
Time Frame: Mean dietary behaviour score as measured by the overall DHQ score, 1 month after the end of the behavioural weight loss program
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Overall score on DHQ
Arm/Group | Motivational Interviewing | Attention Control
Number analyzed (Participants) | 60 | 52
Overall score on DHQ | 2.71 (.04) | 2.67 (.04)
Statistical Analysis 1: Comparison: Motivational Interviewing vs Attention Control; Linear Mixed Modelling (LMM) was used; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p > .05, Mixed Models Analysis — Significance threshold is p=.05

11. Secondary Outcome: Dietary Behaviour at 6 Month Follow up
Description: as for outcome 9
Time Frame: Mean dietary behaviour score as measured by the overall DHQ score, 6 months after the end of the behavioural weight loss program
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Overall score on DHQ
Arm/Group | Motivational Interviewing | Attention Control
Number analyzed (Participants) | 60 | 56
Overall score on DHQ | 2.80 (.04) | 2.70 (.04)
Statistical Analysis 1: Comparison: Motivational Interviewing vs Attention Control; Linear Mixed Modelling (LMM) was used; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p > .05, Mixed Models Analysis — Significance threshold is p=.05

12. Secondary Outcome: Blood Pressure at End of the Behavioural Weight Loss Program, Week 12
Description: A measure of systolic and diastolic blood pressure was taken in a standardized manner according to the Canadian Hypertension Education Program Guidelines (Hemmelgarn et al., 2006). Three different readings of blood pressure were taken at each time point (baseline and end of behavioural weight loss program), and the average of the three readings was taken as the measure of blood pressure for each time point.
Time Frame: Mean blood pressure at the end of the behavioural weight loss program (week 12)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Motivational Interviewing | Attention Control
Number analyzed (Participants) | 64 | 64
mmHg
  Systolic blood pressure | 127.84 (1.03) | 127.19 (1.05)
  Diastolic blood pressure | 77.48 (.68) | 77.89 (.68)
Statistical Analysis 1: Comparison: Motivational Interviewing vs Attention Control; Linear Mixed Modelling (LMM) was used; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p > .05, Mixed Models Analysis — Significance threshold is p=.05

13. Secondary Outcome: Blood Pressure at 6 Month Follow up
Description: A measure of systolic and diastolic blood pressure was taken in a standardized manner according to the Canadian Hypertension Education Program Guidelines (Hemmelgarn et al., 2006). Three different readings of blood pressure were taken at each time point (baseline and 6 month follow up), and the average of the three readings was taken as the measure of blood pressure for each time point.
Time Frame: Mean blood pressure 6 months after the end of the behavioural weight loss program
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Motivational Interviewing | Attention Control
Number analyzed (Participants) | 64 | 56
mmHg
  Systolic blood pressure | 128.93 (1.03) | 128.67 (1.09)
  Diastolic blood pressure | 76.77 (.69) | 77.82 (.72)
Statistical Analysis 1: Comparison: Motivational Interviewing vs Attention Control; Linear Mixed Modelling (LMM) was used; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p > .05, Mixed Models Analysis — Significance threshold is p=.05

14. Secondary Outcome: Eating Disorder Symptomology at End of the Behavioural Weight Loss Program, Week 12
Description: Eating disorder symptomology was measured using the Eating Disorder Examination-Questionnaire (EDE-Q; Fairburn & Beglin, 1994). This self-report questionnaire assesses the presence and degree of specific psychopathology associated with eating disorders over the previous 28 days. Consists of a global score as well as four subscales: Eating Concern, Restraint, Shape Concern, and Weight Concern. The global score is obtained by summing the subscale scores and then dividing this sum by the number of subscales (i.e. four). Range is 0 - 6. Higher scores are indicative of greater eating disorder symptomatology (i.e., worse outcome).
Time Frame: Mean eating disorder symptomology as measured by the global EDE-Q score, at the end of the behavioural weight loss program (week 12)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Global EDE-Q score
Arm/Group | Motivational Interviewing | Attention Control
Number analyzed (Participants) | 59 | 59
Global EDE-Q score | 2.01 (.08) | 2.07 (.08)
Statistical Analysis 1: Comparison: Motivational Interviewing vs Attention Control; Linear Mixed Modelling (LMM) was used; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p > .05, Mixed Models Analysis — Significance threshold is p=.05

15. Secondary Outcome: Eating Disorder Symptomology at 1 Month Follow up
Description: as for outcome 14
Time Frame: Mean eating disorder symptomology as measured by the global EDE-Q score, 1 month after the end of the behavioural weight loss program
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Global EDE-Q score
Arm/Group | Motivational Interviewing | Attention Control
Number analyzed (Participants) | 59 | 51
Global EDE-Q score | 1.91 (.08) | 2.13 (.09)
Statistical Analysis 1: Comparison: Motivational Interviewing vs Attention Control; Linear Mixed Modelling (LMM) was used; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p > .05, Mixed Models Analysis — Significance threshold is p=.05

16. Secondary Outcome: Eating Disorder Symptomology at 6 Month Follow up
Description: as for outcome 14
Time Frame: Mean eating disorder symptomology as measured by the global EDE-Q score, 6 months after the end of the behavioural weight loss program
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Global EDE-Q score
Arm/Group | Motivational Interviewing | Attention Control
Number analyzed (Participants) | 58 | 55
Global EDE-Q score | 1.96 (.08) | 1.92 (.08)
Statistical Analysis 1: Comparison: Motivational Interviewing vs Attention Control; Linear Mixed Modelling (LMM) was used; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p > .05, Mixed Models Analysis — Significance threshold is p=.05

17. Secondary Outcome: Self-efficacy Related to Eating Patterns After the First Motivational Interviewing or Attention Control Interview, Week 1 - 2
Description: Self-efficacy related to eating patterns was measured by the Weight Efficacy Life-Style Questionnaire (WEL; Clark, Abrams, Niaura, Eaton, & Rossi, 1991). This self-report questionnaire yields five subscale scores, which rate self-efficacy for controlling eating in different situations/dimensions: negative emotions, availability, social pressure, physical discomfort, and positive activities. A global/total score (which ranges from 0 - 180) is obtained by summing the scores of each of the five subscales. Higher scores are indicative of greater self-efficacy (i.e., higher scores = better outcome).
Time Frame: Mean self-efficacy related to eating patterns measured immediately after the first MI or attention control interview (week 1 to 2)
Measure: Mean (Standard Deviation); unit: Global score on WEL
Arm/Group | Motivational Interviewing | Attention Control
Number analyzed (Participants) | 69 | 66
Global score on WEL | 136.71 (23.79) | 130.71 (23.79)
Statistical Analysis 1: Comparison: Motivational Interviewing vs Attention Control; Self-efficacy was analyzed via an independent sample t-test comparing the groups on mean global self efficacy rating on the WEL; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; p > .05, t-test, 2 sided — Significance threshold is p=.05

18. Secondary Outcome: Self-efficacy for Engaging in Physical Activity After the First Motivational Interviewing or Attention Control Interview, Week 1- 2
Description: Self-efficacy for engaging in physical activity was measured by the Exercise Self-Efficacy questionnaire (ESE; Nigg & Riebe, 2002). Participants rate their confidence that they could exercise on a 5-point Likert scale for six barriers to exercise (e.g., bad weather, stress, availability of equipment). Consists of a global score as well as four subscales: Eating Concern, Restraint, Shape Concern, and Weight Concern. The global score is obtained by summing the subscale scores and then dividing this sum by the number of subscales (i.e. four). Range is 0 - 6. Higher scores are indicative of greater eating disorder symptomatology (i.e., worse outcome).
Time Frame: Mean self-efficacy for engaging in physical activity measured immediately after the first MI or attention control interview (week 1 - 2)
Measure: Mean (Standard Deviation); unit: ESE score
Arm/Group | Motivational Interviewing | Attention Control
Number analyzed (Participants) | 69 | 66
ESE score | 3.28 (.75) | 3.05 (.81)
Statistical Analysis 1: Comparison: Motivational Interviewing vs Attention Control; Self-efficacy was analyzed via an independent sample t-test comparing the groups on mean self efficacy rating on the ESE; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; p > .05, t-test, 2 sided — Significance threshold is p=.05

19. Secondary Outcome: Self-efficacy Related to Eating Patterns After the Second Motivational Interviewing or Attention Control Interview, Week 12
Description: as for outcome 17
Time Frame: Mean self-efficacy related to eating patterns measured immediately after the second MI or attention control interview (week 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Global score on WEL
Arm/Group | Motivational Interviewing | Attention Control
Number analyzed (Participants) | 67 | 62
Global score on WEL | 148.46 (20.98) | 147.44 (20.75)
Statistical Analysis 1: Comparison: Motivational Interviewing vs Attention Control; [analysis description as in outcome 17, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; p > .05, t-test, 2 sided — Significance threshold is p=.05

20. Secondary Outcome: Self-efficacy for Engaging in Physical Activity After the Second Motivational Interviewing or Attention Control Interview, Week 12
Description: as for outcome 18
Time Frame: Mean self-efficacy for engaging in physical activity measured immediately after the second MI or attention control interview (week 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ESE score
Arm/Group | Motivational Interviewing | Attention Control
Number analyzed (Participants) | 67 | 62
ESE score | 3.58 (.65) | 3.49 (.83)
Statistical Analysis 1: Comparison: Motivational Interviewing vs Attention Control; [analysis description as in outcome 18, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; p > .05, t-test, 2 sided — Significance threshold is p=.05

21. Secondary Outcome: Importance of Change Ratings After the First Motivational Interview or Attention Control Interview, Week 1 - 2
Description: Self-report ratings of "importance of change" after the first motivational interview or attention control interview, on 11-point visual analogue scales (Miller & Rollnick, 2002). For the visual analogue scales, participants were asked to rate how important it is for them personally to lose weight on a scale from 0 "not important" to 10 was "very important". Thus lower scores reflect lower levels of importance for change, and higher scores reflect higher levels of importance for change. Their raw score from 0 to 10 on this measure was taken as their "Importance for Change" rating score.
Time Frame: Importance of change ratings measured immediately after the first MI or attention control interview (week 1- 2)
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Motivational Interviewing | Attention Control
Number analyzed (Participants) | 69 | 66
scores on a scale | 8.67 (1.30) | 8.73 (1.60)
Statistical Analysis 1: Comparison: Motivational Interviewing vs Attention Control; Importance of Change ratings were analyzed via an independent sample t-test comparing the groups on mean Importance of Change ratings on the 11-point visual analogue scales; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; p > .05, t-test, 2 sided — Significance threshold is p=.05

22. Secondary Outcome: Readiness for Change Ratings After the First Motivational Interview or Attention Control Interview, Week 1 -2
Description: Self-report ratings of "readiness for change" after the first motivational interview or attention control interview, on 11-point visual analogue scales (Miller & Rollnick, 2002). For the visual analogue scales, participants were asked to rate how ready they are to lose weight on a scale from 0 "not ready" to 10 was "very ready". Thus lower scores reflect lower levels of readiness for change, and higher scores reflect higher levels of readiness for change. Their raw score from 0 to 10 on this measure was taken as their "Readiness for Change" rating score.
Time Frame: Readiness for change ratings measured immediately after the first MI or attention control interview (week 1- 2)
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Motivational Interviewing | Attention Control
Number analyzed (Participants) | 69 | 66
scores on a scale | 8.64 (1.32) | 8.65 (1.22)
Statistical Analysis 1: Comparison: Motivational Interviewing vs Attention Control; Readiness for Change ratings were analyzed via an independent sample t-test comparing the groups on mean Readiness for Change ratings on the 11-point visual analogue scales; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; p > .05, t-test, 2 sided — Significance threshold is p=.05

23. Secondary Outcome: Confidence for Change Ratings After the First Motivational Interview or Attention Control Interview, Week 1- 2
Description: Self-report ratings of "confidence for change" after the first motivational interview or attention control interview, on 11-point visual analogue scales (Miller & Rollnick, 2002). For the visual analogue scales, participants were asked to rate how confident they feel about succeeding with losing weight on a scale from 0 "not confident" to 10 was "very confident". Thus lower scores reflect lower levels of confidence for change, and higher scores reflect higher levels of confidence for change. Their raw score from 0 to 10 on this measure was taken as their "Confidence for Change" rating score.
Time Frame: Confidence for change ratings measured immediately after the first MI or attention control interview (week 1- 2)
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Motivational Interviewing | Attention Control
Number analyzed (Participants) | 69 | 66
scores on a scale | 7.85 (1.54) | 8.06 (1.38)
Statistical Analysis 1: Comparison: Motivational Interviewing vs Attention Control; Confidence for Change ratings were analyzed via an independent sample t-test comparing the groups on mean Confidence for Change ratings on the 11-point visual analogue scales; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; p > .05, t-test, 2 sided — Significance threshold is p=.05

24. Secondary Outcome: Importance for Change Ratings After the Second Motivational Interview or Attention Control Interview, Week 12
Description: Self-report ratings of "importance of change" after the second motivational interview or attention control interview, on 11-point visual analogue scales (Miller & Rollnick, 2002). For the visual analogue scales, participants were asked to rate how important it is for them personally to lose weight on a scale from 0 "not important" to 10 was "very important". Thus lower scores reflect lower levels of importance for change, and higher scores reflect higher levels of importance for change. Their raw score from 0 to 10 on this measure was taken as their "Importance for Change" rating score.
Time Frame: Importance of change ratings measured immediately after the second MI or attention control interview (week 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Motivational Interviewing | Attention Control
Number analyzed (Participants) | 67 | 62
scores on a scale | 8.52 (1.23) | 8.88 (1.54)
Statistical Analysis 1: Comparison: Motivational Interviewing vs Attention Control; [analysis description as in outcome 21, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; p > .05, t-test, 2 sided — Significance threshold is p=.05

25. Secondary Outcome: Readiness for Change Ratings After the Second Motivational Interviewing or Attention Control Interview, Week 12
Description: Self-report ratings of "readiness for change" after the second motivational interview or attention control interview, on 11-point visual analogue scales (Miller & Rollnick, 2002). For the visual analogue scales, participants were asked to rate how ready they are to lose weight on a scale from 0 "not ready" to 10 was "very ready". Thus lower scores reflect lower levels of readiness for change, and higher scores reflect higher levels of readiness for change. Their raw score from 0 to 10 on this measure was taken as their "Readiness for Change" rating score.
Time Frame: Readiness for change ratings measured immediately after the second MI or attention control interview (week 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Motivational Interviewing | Attention Control
Number analyzed (Participants) | 67 | 62
scores on a scale | 8.70 (1.14) | 8.86 (1.33)
Statistical Analysis 1: Comparison: Motivational Interviewing vs Attention Control; [analysis description as in outcome 22, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; p > .05, t-test, 2 sided — Significance threshold is p=.05

26. Secondary Outcome: Confidence for Change Ratings After the Second Motivational Interviewing or Attention Control Interview, Week 12
Description: Self-report ratings of "confidence for change" after the second motivational interview or attention control interview, on 11-point visual analogue scales (Miller & Rollnick, 2002). For the visual analogue scales, participants were asked to rate how confident they feel about succeeding with losing weight on a scale from 0 "not confident" to 10 was "very confident". Thus lower scores reflect lower levels of confidence for change, and higher scores reflect higher levels of confidence for change. Their raw score from 0 to 10 on this measure was taken as their "Confidence for Change" rating score.
Time Frame: Confidence for change ratings measured immediately after the second MI or attention control interview (week 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Motivational Interviewing | Attention Control
Number analyzed (Participants) | 67 | 62
scores on a scale | 8.25 (1.20) | 8.39 (1.26)
Statistical Analysis 1: Comparison: Motivational Interviewing vs Attention Control; [analysis description as in outcome 23, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; p > .05, t-test, 2 sided — Significance threshold is p=.05

ADVERSE EVENTS:
Description: Serious and Other [Not Including Serious] Adverse Events were not monitored/assessed.
Arm/Group | Motivational Interviewing | Attention Control
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No